CLINICAL TRIAL: NCT00005285
Title: Effect of Maternal Smoking On Neonatal Lung Function
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2006; R01HL036474 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2001-04

CONDITIONS: Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To determine factors, including maternal cigarette smoking and acute respiratory illness, influencing infant lung function at birth and up to five years of age.

DETAILED DESCRIPTION:
BACKGROUND:

Over the past four decades, a significant research effort has been devoted to the understanding of the epidemiology and pathophysiology of chronic obstructive airways disease (COPD) in adult life. Epidemiologic studies uniformly have identified cigarette smoking as the predominant risk factor for the occurrence of COPD. Other factors such as socioeconomic status, environmental pollution, occupational exposures, and inherent genetic susceptibility have been observed to have very limited roles as risk factors.

A number of studies have suggested that postnatal maternal cigarette smoking has a measurable effect on lung function in children. One longitudinal analysis of this problem in children 5-19 years of ages identified significant effects on the growth of FEV1 and forced expiratory flow between the 25th and 75th percent volume points (FEF25-75) of the volume-time curve. These investigators, however, pointed out that the effects which they observed could have resulted from the in utero consequences of maternal smoking during pregnancy and/or from exposure to factors such as severe respiratory illnesses which have been documented to occur with increased frequency early in infancy and were not measured by the study.

DESIGN NARRATIVE:

Pregnant women were identified during the first trimester and followed monthly. Assessments were made of their smoking habits, urinary cotinine measurements, general medical condition, and status of pregnancy. Within two weeks of birth the infants were evaluated with partial forced expiratory flow-volume curves and measurement of passive respiratory system compliance and resistance. Measurements were repeated at intervals until age five. Babies were also observed regularly for respiratory illness experience, passive exposure to cigarette smoke, and general respiratory health.

The study helped to elucidate: the effect of maternal cigarette smoking on lung function at birth and development of function at five years; the effects of postnatal factors on lung development; the extent to which the reported increased frequency of respiratory illness in infants of smoking mothers resulted from in utero exposure to tobacco smoke products or postnatal passive smoking.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-07; Study Completion 1996-11 (Actual)

REFERENCES:
- [Background] David MM, Hanrahan JP, Carey V, Speizer FE, Tager IB. Respiratory symptoms in urban Hispanic and non-Hispanic white women. Am J Respir Crit Care Med. 1996 Apr;153(4 Pt 1):1285-91. doi: 10.1164/ajrccm.153.4.8616555.
- [Background] Weiss ST, Ware JH. Overview of issues in the longitudinal analysis of respiratory data. Am J Respir Crit Care Med. 1996 Dec;154(6 Pt 2):S208-11. doi: 10.1164/ajrccm/154.6_Pt_2.S208. No abstract available. PMID 8970389
- [Background] Rijcken B, Weiss ST. Longitudinal analyses of airway responsiveness and pulmonary function decline. Am J Respir Crit Care Med. 1996 Dec;154(6 Pt 2):S246-9. doi: 10.1164/ajrccm/154.6_Pt_2.S246. No abstract available. PMID 8970396
- [Background] Hanrahan JP, Segal MR, Chervin BS, Barr MB, VanVunakis H, Weiss ST, Speizer FE, Tager IB: Early vs. Late Prenatal Smoking: Effect on Birth Rate. Am Rev Respir Dis, 137:253, 1988
- [Background] Chervin BS, Barr MB, Hanrahan JP, Segal MR, VanVunakis H, Weiss ST, Tager IB, Speizer FE: Assessment of Prenatal Infant Exposure to Maternal Smoking. Am Rev Respir Dis, 137:253, 1988
- [Background] Hanrahan JP, Castile RG, Segal MR, Aylward D, Barr MB, Chervin BS, Tager IB, Speizer FE, Weiss ST: Longitudinal Lung and Airway Growth in Healthy Infants in the First 6 Months of Life. Am Rev Respir Dis, 137:381, 1988
- [Background] Hanrahan JP, Tager IB, Castile RG, Segal MR, Weiss ST, Speizer FE. Pulmonary function measures in healthy infants. Variability and size correction. Am Rev Respir Dis. 1990 May;141(5 Pt 1):1127-35. doi: 10.1164/ajrccm/141.5_Pt_1.1127. PMID 2339835
- [Background] Hanrahan JP, Tager IB, Segal MR, Tosteson TD, Castile RG, Van Vunakis H, Weiss ST, Speizer FE. The effect of maternal smoking during pregnancy on early infant lung function. Am Rev Respir Dis. 1992 May;145(5):1129-35. doi: 10.1164/ajrccm/145.5.1129. PMID 1586058
- [Background] Weiss ST. Problems in the phenotypic assessment of asthma. Clin Exp Allergy. 1995 Nov;25 Suppl 2:12-4; discussion 17-8. doi: 10.1111/j.1365-2222.1995.tb00410.x. No abstract available. PMID 8590331
- [Background] Adler A, Tager IB, Brown RW, Ngo L, Hanrahan JP. Relationship between an index of tidal flow and lower respiratory illness in the first year of life. Pediatr Pulmonol. 1995 Sep;20(3):137-44. doi: 10.1002/ppul.1950200303. PMID 8545164
- [Background] Brown RW, Hanrahan JP, Castile RG, Tager IB. Effect of maternal smoking during pregnancy on passive respiratory mechanics in early infancy. Pediatr Pulmonol. 1995 Jan;19(1):23-8. doi: 10.1002/ppul.1950190105. PMID 7675554
- [Background] Tager IB, Hanrahan JP, Tosteson TD, Castile RG, Brown RW, Weiss ST, Speizer FE. Lung function, pre- and post-natal smoke exposure, and wheezing in the first year of life. Am Rev Respir Dis. 1993 Apr;147(4):811-7. doi: 10.1164/ajrccm/147.4.811. PMID 8466114
- [Background] Tager IB, Ngo L, Hanrahan JP. Maternal smoking during pregnancy. Effects on lung function during the first 18 months of life. Am J Respir Crit Care Med. 1995 Sep;152(3):977-83. doi: 10.1164/ajrccm.152.3.7663813.